CLINICAL TRIAL: NCT04216251
Title: PREPARE: PRevention Using EPA Against coloREctal Cancer
Brief Title: PRevention Using EPA Against coloREctal Cancer
Acronym: PREPARE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mingyang Song, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-402; NCT04172636 (obsolete NCT alias)
Record Dates: First submitted 2019-12-19; First posted 2020-01-02 (Actual); Results first posted 2024-02-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Adenoma; Colorectal Cancer; Endoscopic Surgery; Eicosapentaenoic Acid; Gastrointestinal Microbiome
Keywords: Colorectal Adenoma; Colorectal Cancer; colonoscopic Surgery; Endoscopic Surgery; Eicosapentaenoic acid; Gastrointestinal Microbiome; Mucosal Tissue
MeSH Terms: conditions — Colorectal Neoplasms | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMR101 (Experimental): Study procedures include screening for eligibility and study treatment including ARM101 Lifestyle questionnaire, Nutritional survey. Flexible sigmoidoscopy (24 biopsies of normal colorectal mucosa, one stool sample),blood, evaluations, and follow up visits.
  - AMR101-oral predetermined protocol dosage, daily for a minimum of 8 weeks and maximum of 12 weeks
  Interventions: Drug: AMR101

INTERVENTIONS:
Drug: AMR101 — AMR101-oral predetermined protocol dosage, daily for a minimum of 8 weeks and maximum of 12 weeks
  Other Names: VASCEPA

SUMMARY:
This research study is evaluating the effect of AMR101 as a possible chemopreventive agent to reduce risk of colorectal cancer in individuals with a history of colorectal adenoma.

- The name of the study drug involved in this study is:

-- AMR101 (VASCEPA).

DETAILED DESCRIPTION:
This prospective, single-arm, research study evaluating the effect of AMR101, as a chemopreventive agent to reduce risk of colorectal cancer in individuals with a history of colorectal adenoma.

* AMR101 is made of marine omega-3 fatty acid, which is a family of natural substances found in the oil of certain fish, such as salmon and mackerel. Marine omega-3 fatty acid cannot be produced in sufficient amount by the human body and has to be obtained through diet or supplemented to maintain normal function in the body.
* The U.S. Food and Drug Administration (FDA) has not approved AMR101 as a treatment for any disease.
* AMR101 is commercially available in the US as VASCEPA (icosapent ethyl)
* The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits, including:

  * Lifestyle questionnaire,
  * Nutritional survey
  * Flexible sigmoidoscopy (24 biopsies of normal colorectal mucosa, one stool sample)
  * Blood samples,
* AMR101 administered daily, orally for 8-12 weeks and it is expected 80 participants will take part.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Underwent screening or surveillance colonoscopy with removal of at least one adenoma;
* Age 18-80 years.

  * This study will only include adult participants because colorectal carcinogenesis in children is more likely to be related to a cancer predisposition syndrome with distinct biological mechanisms compared with sporadic colorectal cancer in adults. Patients over age 80 will not be enrolled since the benefits and risks of AMR101 over the age of 80 have not yet been well-characterized.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* The effects of AMR101 on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Subjects must be able and willing to follow study procedures and instructions.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study

* Currently using or have used any fish oil supplement at any dose more than once per week within the last month
* Regularly consuming more than three servings of fish per week.
* History of allergic reactions attributed to fish or compounds of similar chemical or biologic composition to omega-3 fatty acid.
* Diagnosis of inflammatory bowel disease, liver or kidney disease, bleeding diathesis
* Any prior diagnosis of gastrointestinal cancer (including esophageal, small intestine, colon, pancreatic), or any diagnosis of other cancers (with the exception of nonmelanoma skin) in which there has been any active treatment within the last three years.
* Known diagnosis of Familial Adenomatous Polyposis (FAP) or Hereditary Non-Polyposis Colorectal Cancer (HNPCC, Lynch Syndrome).
* Any adenoma that was not completely removed during previous colonoscopy.
* Known bleeding tendency/condition (e.g. von Willebrand disease) or history of peptic ulcer or gastrointestinal bleed, endoscopic complications, or contraindication to colonoscopy.
* Current use of anticoagulant therapies, including Heparin, Warfarin, Dalteparin sodium,Bivalirudin, Argatroban, Lepirudin, Heparin Sodium, Heparin/Dextrose, and an unwillingness or inability to discontinue anticoagulants.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inability or unwillingness to abstain from non-protocol use of fish oil supplements or to provide blood or stool samples or colon biopsies during the study.
* Participants who are receiving any other investigational agents.
* Inability or unwillingness to swallow pills.
* Pregnant or breastfeeding. The effects of AMR101 on the developing human fetus are unknown. For this reason,women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Similarly, lactating women are excluded from this study because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with AMR101. Consequently, breastfeeding should be discontinued if the mother is enrolled on the study.
* Known positive test for human immunodeficiency virus (HIV), hepatitis C virus, or acute or chronic hepatitis B infection. Participants with these infections are ineligible because they are at increased risk of significant complications in the perioperative period, and because fresh tissue from patients with these infections cannot be harvested for research purposes, per institutional policy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mingyang Song, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who meet the inclusion criteria will be identified through investigators during their routine clinical practice, supplemented by a periodic query of the MGH endoscopy and pathology databases. Potentially eligible participants are approached by letter from their treating physician. Two weeks after receiving the letter, study staff will contact eligible parties and screen for eligibility via phone interview. Enrollment began in December 2020 and ended in September 2022.
Groups:
- AMR101: The first dose of the study medication will be given to patients after the initial flexible sigmoidoscopy. Participants will be expected to take 4 0.5 gram capsules orally, twice daily (daily dose of 4 grams) for a minimum of 8 weeks and maximum of 12 weeks
Period: Overall Study
Arm/Group | AMR101
Started | 81
Completed | 73
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: We have enrolled 81 healthy participants between the ages of 18 and 80 who have undergone screening or surveillance colonoscopy with removal of at least one adenoma and was not regularly using fish oil supplements or consuming more than 3 servings of fish per week.
Arm/Group | AMR101
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.95 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 76
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in the Marine Omega-3 Polyunsaturated Fatty Acid (MO3PUFA) Composition in Colorectal Tissues as a Result of the AMR101 Treatment.
Description: Measured using the extraction of fatty acid with gas chromatography-mass spectrometry from the biopsy tissue.
Time Frame: 8-12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total fatty acids
Groups:
- Pre-treatment: This is the baseline (e.g., pre-treatment) measurement.
- Post-treatment: This is the post-treatment measurement.
Arm/Group | Pre-treatment | Post-treatment
Number analyzed (Participants) | 59 | 59
percentage of total fatty acids | 0.54 (0.33) | 2.95 (1.65)

2. Secondary Outcome: Change in the Gut Microbiome Composition
Description: Measured using shotgun metagenomic sequencing of microbial DNA on pre- and post-treatment stool samples.
  The reported results represent the Shannon Diversity Index, which is a quantitative measure that reflects how many different bacterial species there are in a sample. The index's values range from 0 to 5, but usually range from 1.5 to 3.5. The greater the index, the more diverse the gut microbiota. A negative change indicates a decrease in diversity and a positive change indicates an increase in diversity.
  We used the vegan R package to conduct the analysis.
Time Frame: 8-12 weeks 8-12 weeks 8-12 weeks 8-12 weeks
Population: This is after quality control filtering and excluding participants who had missing pre- or post-treatment samples.
Measure: Median (Inter-Quartile Range); unit: Shannon diversity index
Arm/Group | Pre-treatment | Post-treatment
Number analyzed (Participants) | 67 | 67
Shannon diversity index | 3.082 [2.927 to 3.266] | 3.133 [2.968 to 3.281]

3. Secondary Outcome: Change in Fecal Metabolite Levels (Butyrate)
Description: Butyrate is the metabolite of our most interest for the current study, based on the prior data suggesting that marine omega-3 fatty acid may increase the production of butyrate by bacterial fermentation of dietary fiber.
  The metabolites were measured by the non-targeted global metabolomic panel. The measurement represents the abundance (assessed as weight percentage of density) of a metabolite after total-signal normalization to account for varying water weight across stool samples.
Time Frame: 8-12 weeks
Population: This is after quality control filtering and excluding participants who had missing pre- or post-treatment samples.
Measure: Median (Inter-Quartile Range); unit: Weight percentage of butyrate density
Arm/Group | Pre-treatment | Post-treatment
Number analyzed (Participants) | 64 | 64
Weight percentage of butyrate density | 0.64 [0.42 to 0.81] | 0.63 [0.39 to 0.76]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | AMR101
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 1/81
Other Adverse Events (participants affected / at risk) | 20/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMR101 (N=81)
Ischemic right foot with thrombosis of right external iliac artery stent and common femoral artery (Vascular disorders) | 1 — Peripheral ischemia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMR101 (N=81)
GI Upset (i.e. nausea/gas/diarrhea/constipation/stomach ache/loss of appetite) (Gastrointestinal disorders) | 12
COVID and Flu-like symptoms (congestion, chills, fever, body ache, headache) (Infections and infestations) | 4
Chest pain (Respiratory, thoracic and mediastinal disorders) | 2
Skin issues (acne, hyperpigmentation) (Skin and subcutaneous tissue disorders) | 2
Pain (joint pain, muscle aches) (Musculoskeletal and connective tissue disorders) | 3
Esophagitis (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT04216251/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04216251/ICF_001.pdf